CLINICAL TRIAL: NCT04588766
Title: Evaluation of Posture, Sleep, Physical Activity and Quality of Life in Individuals With Chronic Constipation With Cerebral Palsy
Brief Title: Chronic Constipation With Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Şeyma Nur Önal, Lecturer, Bartın Unıversity
Other Study IDs: constipationandcerebralpalsy
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Constipation; Physical activity; Posture; Quality of life; Sleep
MeSH Terms: conditions — Cerebral Palsy; Constipation; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- constipation group: Constipation symptoms of individuals with cerebral palsy who were randomly evaluated were questioned and recorded according to Rome IV criteria. The group with cerebral palsy constipation was included in this group.
  Interventions: Other: constipation group
- control group: Constipation symptoms of individuals with cerebral palsy who were evaluated randomly were questioned and recorded according to Rome IV criteria. The group with cerebral palsy without constipation was included in this group.
  Interventions: Other: control group

INTERVENTIONS:
Other: constipation group — Constipation symptoms of individuals with cerebral palsy who were randomly evaluated were questioned and recorded according to Rome IV criteria. The group with cerebral palsy constipation was included in this group.
  Groups: constipation group
Other: control group — Constipation symptoms of individuals with cerebral palsy who were evaluated randomly were questioned and recorded according to Rome IV criteria. The group with cerebral palsy without constipation was included in this group.
  Groups: control group

SUMMARY:
This study was performed to evaluate posture, sleep, physical activity and quality of life in individuals with chronic constipation Cerebral Palsy.

DETAILED DESCRIPTION:
The study included 81 individuals diagnosed with CP, 3-18 years of age and 2 groups with and without constipation according to Rome IV criteria.

General motor impairment levels with "Gross Motor Function Classification System, motor functions with "Gross Motor Function Measurement, functional independence levels Functional Independence Measurement, spasticity Modified Ashworth Scale , posture characteristics Spinal Aligment and Range of Motion Measurement, with stool characteristics Bristol Stool Form Scale the presence and severity of constipation with the Modified Constipation Assessment Scale and Constipation Severity Scale sleep quality with Pediatric Sleep Questionnaire physical activity level Physical Activity Scale and life quality was evaluated with Pediatric Quality of Life Inventory .

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Being between the ages of 2-18
* Being diagnosed with Cerebral Palsy

Exclusion Criteria:

* • Having undergone surgery involving intestinal health
* Having a chronic infectious bowel disease
* Having a congenital bowel anomaly
* Having received botox treatment in the last six months

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study included 81 individuals diagnosed with CP, 3-18 years of age and 2 groups with and without constipation according to Rome IV criteria.
Sampling Method: Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Bristol poop scale | 5 minutes
  The Bristol Poop Scale is a 7-point scale and was used to define stool consistency. It has been shown that the Bristol Poop Scale is associated with constipation and colonic transit time in children without constipation (140). Hard stools fit 1 and 2, loose (ideal) stools fit 3, 4, 5, diarrhea types 6 and 7. Therefore, represented by stool consistency scores as hard, loose stools and diarrhea.

SECONDARY OUTCOMES:
Gross motor function criterion | 20 minutes
  The Gross Motor Function Scale-88 was created to evaluate the changes in gross motor functions as growth and development continues in individuals with cerebral palsy. It is a standardized, regular, systematic observational test. It has categories that follow each other during normal motor and physiological development. These; are supine, prone, crawling, sitting, laptop, standing, walking, and use of stairs. These categories include activities appropriate to the headings in the sub-items. Scoring is divided into five main categories. It consists of a total of 88 items, 17 in the supine and prone categories, 20 in the sitting category, 14 in the crawling and laptop category, 13 in the standing category, and 24 in the walking, running and stair climbing categories. While these items are tested, gross motor functions are evaluated according to the correct achievement level.
The Gross Motor Function Classification System | 2 minutes
  The Gross Motor Function Classification System was used to classify the gross motor function levels of individuals with CP. This system is a standard classification system developed by Robert Palisano. KMFSS is based on actively initiated movements by the individual, focusing on sitting, position change and mobility. In this five-level system, it is important that the differences between levels are evident in life activities. The differences are determined by the limitations in functional activities, the need for manual movement aids (walkers, canes, crutches, etc.) or wheeled transport vehicles. The quality of the movement is of little importance
Rome IV criteria | 5
  Constipation is not a disease but a symptom. Constipation is determined according to Rome IV criteria. Symptoms should have started at least 6 months ago. At least 25% of the defecations; in the form of lumpy or hard stools, straining, feeling of anorectal obstruction, feeling of incomplete emptying, using hand aid (finger emptying effort, pelvic floor support); The frequency of defecation should include two or more of the findings of defecation less than 3 times a week, soft stools if laxative is not used, very rare, and not having sufficient criteria for the diagnosis of inflammatory bowel syndrome. The identified complaints must continue for at least 3 months.
Modified constipation assessment scale | 5 minutes
  This scale, which will be used to evaluate constipation in individuals, was used in 1989 in McMillan SC. et al. It is a valid and reliable scale consisting of 9 questions that can be answered by the individual about the presence and severity of constipation and can be used in children and adults. It contains eight items, each classified as "no problem" by the patient. It is scored as 'no problem' (0 point), 'some problem' (1 point) or 'serious problem' (2 points). The item scores are then added up and the total score ranges from 0 (no constipation) to 18 (worst possible constipation).
Constipation severity scale | 5 minutes
  To measure the severity of constipation, Varma MG. et al. developed by. CSO is a scale that questions the frequency and intensity of defecation of individuals and the difficulty in this process. This scale, which can provide information about constipation symptoms, consists of 16 questions.
Six-sided pain scale-6 | 2 minutes
  The Hexagonal Pain Scale (YAS-6) was originally developed for use in pediatrics. There are several versions of YAS, some of them six, seven or nine hundred. At the same time, the scale with eleven faces is used in current studies to be compatible with the 0--10 Numeric Rating Scale.
Beverage consumption frequency form | 10 minutes
  Turkish validity for measuring the daily fluid intake in individuals Eda Köksal et al. Beverage Consumption Frequency Form prepared by The Beverage Consumption Frequency Form was adapted from Hedrick and the latest version was created with the most and most frequently consumed beverages in Turkish society.
Sleep form in children | 5 minutes
  This form, prepared to evaluate the sleep conditions of children, was used by Ronald Chervin et al. to assess sleep-related problems in children aged 2-18 years
Physical activity scale | 10 minutes
  The Physical Activity Scale of Preschool Children Dwyer et al. It is a 3-day activity scale developed by
Spinal straightness and normal joint motion | 5 minutes
  Validity in the evaluation of spinal smoothness and general joint mobility in cases Chen, C.L. et al. The Spinal Alignment and Range of Motion Measure (SAROMM) scale made by
Quality of life scale for children | 5 minutes
  The Children's Quality of Life Scale (PedsQL) was used by Varni et al. To measure the health-related quality of life of individuals aged between 2 and 18 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)